CLINICAL TRIAL: NCT05486949
Title: A Phase 1, Single-Center, Nonrandomized, Open-Label, 2-Part, Fixed-Sequence, Drug-Drug Interaction Study to Assess the Pharmacokinetics and Safety of AZD4205 When Orally Administered Alone, When Coadministered With Itraconazole, and When Coadministered With Carbamazepine in Healthy Adult Subjects
Brief Title: Drug-drug Interactions Between AZD4205 and Itraconazole/Carbamazepine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: DZ2021J0002
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Carbamazepine; Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD4205 and carbamazepine (Experimental): Subjects in arm 1 will receive AZD4205 single dose on Day 1, and the second dose of AZD4205 along with carbamazepine after the wash-out period.
  Interventions: Drug: AZD4205 and carbamazepine
- AZD4205 and itraconazole (Experimental): Subjects in arm 2 will receive AZD4205 single dose on Day 1, and the second dose of AZD4205 along with itraconazole after the wash-out period.
  Interventions: Drug: AZD4205 and itraconazole

INTERVENTIONS:
Drug: AZD4205 and carbamazepine — All subjects will receive AZD4205 single dose on Day 1, and the second dose of AZD4205 along with carbamazepine after the wash-out period.
  Arms: AZD4205 and carbamazepine
Drug: AZD4205 and itraconazole — All subjects will receive AZD4205 single dose on Day 1, and the second dose of AZD4205 along with itraconazole after the wash-out period.
  Arms: AZD4205 and itraconazole

SUMMARY:
This is a Phase 1, single-center, nonrandomized, open-label, 2-part, fixed-sequence, drug-drug interaction (DDI) study to assess the effect of multiple doses of itraconazole, a CYP3A4 enzyme inhibitor, on the single dose PK of AZD4205 in healthy adult subjects (Part A) and to assess the effect of multiple doses of carbamazepine, a CYP3A4 inducer, on the single dose PK of AZD4205 in healthy adult subjects (Part B).

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study, give written informed consent, and comply with the study restrictions.
2. Sex: male or female; females may be of childbearing potential, of nonchildbearing potential, or postmenopausal.
3. Age: 18 to 55 years, inclusive, at screening.
4. Body mass index (BMI): 18.0 to 30.0 kg/m2, inclusive, at screening.
5. Weight: ≥55 kg for males and ≥45 kg for females at screening.
6. Status: healthy subjects.
7. Healthy status as defined by the absence of evidence of any clinically significant, in the opinion of the investigator, active, or chronic disease.
8. Ability and willingness to abstain from alcohol-, caffeine-, and methylxanthine containing beverages or food from 72 hours (3 days) prior to admission until discharge from the clinical facility.
9. No clinically significant hematological or coagulation abnormalities, as judged by the investigator.
10. Male subjects and female subjects of childbearing potential must agree to use protocol specified methods of contraception and comply with pregnancy precautions as described in the protocol.
11. All prescription medications must have been stopped at least 28 days or 5 half lives, if known prior to the admission to the clinical research center.
12. All over the counter medication must have been stopped at least 14 days or 5 half-lives, prior to the admission to the clinical research center.
13. Normal baseline ECG (QTcF <450 msec, PR <220 msec).
14. Adequate organ function, defined by the absence of any clinically significant abnormalities, as judged by the investigator, of the relevant baseline clinical safety assessments.

Exclusion Criteria:

1. Employee of PRA or the sponsor.
2. Any condition which, in the opinion of the investigator, would interfere with the subject's ability to provide informed consent, comply with study instructions, confound interpretation of study results, or endanger the subject if he or she takes part in the trial.
3. Women who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 30 days after the last dose of study drug.
4. For all females of childbearing potential: positive pregnancy test at screening or at admission to the clinic.
5. Males with female partners who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 90 days after the last dose of study drug.
6. Use of any investigational drug or device within 30 days, or investigational biologics within 120 days before the first dose of study drug.
7. Any disease which, in the opinion of the investigator, poses an unacceptable risk to the subject.
8. Clinically relevant issues of visual function as determined from the medical history and physical exams, as judged by the investigator.
9. Clinically significant history of any drug sensitivity, drug allergy, or food allergy, as determined by the investigator.
10. History of allergy or hypersensitivity to AZD4205, or other drugs similar in class or similar in chemical structure to AZD4205, as judged by the investigator.
11. History of major surgery or blood transfusion within 30 days prior to the first drug administration.
12. History of malignancy of any type.
13. Evidence of clinically significant or relevant renal, hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
14. Manifestation of malabsorption due to prior gastrointestinal surgery, gastrointestinal disease, or any other reason that may affect the absorption of AZD4205.
15. Positive result from a COVID-19 test per site policy and requirement.
16. Positive test result for alcohol and/or drugs of abuse at screening or on Day -1.
17. Positive test result from Quantiferon-TB Gold test.
18. Presence of pulmonary infections or other clinically significant active infection within 30 days of informed consent.
19. Received COVID-19 vaccine or any live vaccine within 4 weeks prior to the first dose of the investigational medicinal product.
20. Self-reported substance abuse within 12 months of screening.
21. Using tobacco or nicotine products within 90 days prior to the first drug administration.
22. Strenuous activity, sunbathing, and contact sports within 48 hours prior to admission to the clinical facility through follow-up.
23. History of donation of more than 500 mL of blood within 60 days prior to dosing in the clinical research center or planned donation before 30 days has elapsed since intake of study drug.
24. Plasma or platelet donation within 7 days of dosing and through follow-up.
25. History within the previous 12 months of alcohol consumption exceeding 2 standard drinks per day on average.
26. Positive screening test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or HIV 1 and 2 antibodies.
27. Consumption of any nutrients/foods known to modulate CYP450 enzyme activity within 7 days prior to administration of study drug and during the study.
28. Abnormal echocardiogram (ECHO) at baseline, as judged by the investigator.
29. History of allergy, severe adverse reaction, intolerance, or hypersensitivity to itraconazole or other azole antifungals, as determined by the investigator (Part A Only).
30. History of allergy, severe adverse reaction, intolerance, or hypersensitivity to carbamazepine, carboxamide derivatives, or other drugs that are structurally related to carbamazepine, as judged by the investigator (Part B Only).
31. Individuals who have Asian ancestry (including those who have 1 or more Asian grandparent, Part B Only).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of AZD4205 when dosed alone or coadministered with itraconazole (Part A) | up to 10 days after study drug administration when AZD4205 dosed alone; up to 18 days after study drug administration when coadministered with itraconazole
Time to reach maximum plasma concentration (tmax) of AZD4205 when dosed alone or coadministered with itraconazole (Part A) | up to 10 days after study drug administration when AZD4205 dosed alone; up to 18 days after study drug administration when coadministered with itraconazole
Area under the concentration-time curve from time 0 to time of last quantifiable concentration (AUC0-t) when dosed alone or coadministered with itraconazole (Part A) | up to 10 days after study drug administration when AZD4205 dosed alone; up to 18 days after study drug administration when coadministered with itraconazole
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) when dosed alone or coadministered with itraconazole (Part A) | up to 10 days after study drug administration when AZD4205 dosed alone; up to 18 days after study drug administration when coadministered with itraconazole
Maximum plasma concentration (Cmax) of AZD4205 when dosed alone or coadministered with carbamazepine (Part B) | up to 10 days after study drug administration
Time to reach maximum plasma concentration (tmax) of AZD4205 when dosed alone or coadministered with carbamazepine (Part B) | up to 10 days after study drug administration
Area under the concentration-time curve from time 0 to time of last quantifiable concentration (AUC0-t) when dosed alone or coadministered with carbamazepine (Part B) | up to 10 days after study drug administration
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) when dosed alone or coadministered with carbamazepine (Part B) | up to 10 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Shirlian Xu, Study Director — Dizal Pharma
Locations (1):
- Pharmaceutical Research Associates, Inc., Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No